CLINICAL TRIAL: NCT02592369
Title: The Medtronic CoreValve™ Evolut R™ FORWARD Study
Brief Title: CoreValve™ Evolut R™ FORWARD Study
Acronym: FORWARD
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: Evolut R™ FORWARD Study
Record Dates: First submitted 2015-10-20; First posted 2015-10-30 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Medtronic CoreValve™ Evolut R™ System — The Evolut R System is intended for relief of aortic stenosis in patients with symptomatic heart disease due to severe native calcific aortic stenosis who are judged by a heart team, to be at high or extreme risk for open heart surgery. The Evolut R TAV treats aortic stenosis by displacing and functionally replacing the dysfunctional native valve with a bioprosthetic valve delivered on a catheter while the heart is still beating, thus avoiding the risks of cardiopulmonary bypass. Its intended performance is to relieve aortic valve stenosis without inducing significant regurgitation, thereby restoring effective aortic valve function.

SUMMARY:
Prospective, single arm, multi-center, observational, post market study to document the clinical and device performance outcomes of the Evolut R system used in routine hospital practice in a large patient cohort for the treatment of symptomatic native aortic valve stenosis or a stenosed, insufficient, or combined surgical bioprosthetic valve failure necessitating valve replacement.

DETAILED DESCRIPTION:
The study objective is to document the clinical and device performance outcomes of the Evolut R system used in routine hospital practice in a large patient cohort for the treatment of symptomatic native aortic valve stenosis or a stenosed, insufficient, or combined surgical bioprosthetic valve failure necessitating valve replacement.

Prospective, single arm, multi-center, observational, post market study. In Australia and Canada it is a prospective, single arm, multi-center pre-market study.

Up to 60 centers worldwide. Geographies may include Europe, Australia, Middle East and Africa, Latin America and Canada.

Approximately 1000 implanted subjects, consented for follow-up through three years.

For each subject, data will be collected preoperatively, intra-operatively, at hospital discharge, 30 days, 1, 2 and 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic native aortic valve stenosis or a stenosed, insufficient, or combined surgical bioprosthetic valve failure necessitating valve replacement
* Acceptable candidate for elective treatment with the Evolut R System and in conformity with the local regulatory and medico economic context
* Age ≥80 years OR considered to be at high or greater risk for surgical aortic valve replacement (AVR) where high risk is defined as:

  * Society of Thoracic Surgeons (STS) predicted risk of mortality ≥8% OR
  * Documented heart team agreement of risk for AVR due to frailty or comorbidities.
* Geographically stable and willing to return to the implanting site for all follow-up visits
* Of legal age to provide informed consent (patient Informed Consent or Data Release Form) in the country where they enroll in the trial
* The patient has been informed of the nature of the study, is able and willing to provide consent without assistance from a legal representative and has consented to participate, and has authorized the collection and release of his/her medical information by signing a Patient Informed Consent or Data Release Form.

Exclusion Criteria:

* Known hypersensitivity or contraindication to aspirin, heparin (HIT/HITTS) and bivalirudin, ticlopidine, clopidogrel, Nitinol (Titanium or Nickel), or sensitivity to contrast media, which cannot be adequately premedicated
* Preexisting mechanical heart valve in aortic position
* Ongoing sepsis, including active endocarditis
* Anatomically not suitable for the Evolut R system
* Estimated life expectancy of less than 1 year
* Participating in another trial that may influence the outcome of this trial
* Need for emergency surgery for any reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients with symptomatic native aortic valve stenosis or a stenosed, insufficient, or combined surgical bioprosthetic valve failure necessitating valve replacement who are scheduled for an elective transcatheter aortic valve implantation. Patients who will undergo an emergency procedure should not be included in this study.
Sampling Method: Probability Sample
Enrollment: 1060 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
All-cause mortality rate | 30 days post implant
  All-cause mortality rate at 30 days post procedure

SECONDARY OUTCOMES:
Device success according to VARC2 | 24h to 7 days post implant
  Device success rate at 24 hours to 7 days, defined according to the Valve Academic Research Consortium-2 (VARC-2) guidelines as:
  * Absence of procedural mortality, AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location, AND
  * Intended performance of the prosthetic heart valve, defined as the absence of patient-prosthesis mismatch and mean gradient < 20 mmHg (or peak velocity < 3 m/sec), AND No moderate or severe prosthetic valve regurgitation.
Hemodynamic performance | 24h to 7 days and 1 year post implant
  Hemodynamic performance at 24 hours to 7 days (discharge) and 1 year post procedure, including the mean prosthetic valve gradient as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory.
Hemodynamic performance | 24h to 7 days and 1 year post implant
  Hemodynamic performance at 24 hours to 7 days (discharge) and 1 year post procedure, including the effective orifice area as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory.
Hemodynamic performance | 24h to 7 days and 1 year post implant
  Hemodynamic performance at 24 hours to 7 days (discharge) and 1 year post procedure, including the degree of prosthetic valve regurgitation (transvalvular, paravalvular, and total) as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory.
Early safety composite endpoint according to VARC2 | 30 days post implant
  Early Safety composite endpoint at 30 days post procedure, defined according to the VARC-2 guidelines, defined as any of the following components:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury: stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVI, or SAVR)
Event rates according to VARC2 | 30 days post implant
  Event rates of the individual components of the VARC-2 composite Early Safety endpoint at 30 days post procedure
Rate of new permanent pacemaker implant | 30 days post implant
  Rate of new permanent pacemaker implant at 30 days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Grube, Prof. Dr., Principal Investigator — University Hospital, Bonn; Stephan Windecker, Prof. Dr., Principal Investigator — INSELSPITAL, Universitätsspital Bern
Locations (54):
- Australia (4):
  - Flinders Medical Centre, Adelaide
  - Monash Medical Centre, Melbourne
  - The Alfred Hospital, Melbourne
  - Fiona Stanley Hospital Perth, Perth
- Universitair Ziekenhuis Antwerpen, Antwerp, Belgium
- Canada (3):
  - London Health Sciences Centre - University Campus, London
  - Sunnybrook Health Sciences Center, Toronto
  - Saint Paul's Hospital, Vancouver
- Angiografia de Occidente S.A., Cali, Colombia
- Nemocnice Podlesi a.s., Třinec, Czechia
- France (5):
  - Centre Hospitalier Universitaire - Hopital Henri Mondor, Créteil
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Institut Hospitalier Jacques Cartier, Massy
  - Hopital Bichat - Claude Bernard, Paris
  - Clinique Pasteur, Toulouse
- Germany (13):
  - Herz- und Diabeteszentrum NRW - Ruhr-Universitaet Bochum, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - University of Bonn, Cardiology, Bonn
  - Sana-Herzzentrum Cottbus GmbH, Cottbus
  - Herzzentrum Dresden GmbH Universitaetsklinik, Dresden
  - Universitaetsklinikum Düsseldorf, Düsseldorf
  - Elisabeth-Krankenhaus Essen GmbH, Essen
  - Universitätsklinikum Essen, Essen
  - University of Frankfurt, Frankfurt
  - Asklepios Klinik Sankt Georg, Hamburg
  - Städtisches Klinikum Karlsruhe GmbH, Karlsruhe
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum Muenchen - Klinik an der TU Muenchen, Munich
- Hygeia Hospital, Athens, Greece
- Semmelweis Egyetem AOK, Budapest, Hungary
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (5):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Presidio Ospedaliero Ferrarotto Alessi, Catania
  - IRCCS Policlinico San Donato, Milan
  - Ospedale San Raffaele - Milano, Milan
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento di Cisanello, Pisa
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis - Locatie Oosterpark, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
- Oslo Universitetssykehus-Ullevål Universitetssykehus, Oslo, Norway
- Complejo Hospitalario Dr Arnulfo Arias Madrid, Panama City, Panama
- Instytut Kardiologii, Warsaw, Poland
- Centro Hospitalar de Vila Nova de Gaia/Espinho - Unidade I, Vila Nova de Gaia, Portugal
- Prince Sultan Cardiac Center, Riyadh, Saudi Arabia
- Mediclinic Panorama, Cape Town, South Africa
- Spain (3):
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela
- Akademiska Sjukhuset, Uppsala, Sweden
- United Kingdom (4):
  - Royal Victoria Hospital - Belfast Health and Social Care Trust, Belfast
  - Royal Sussex County Hospital, Brighton
  - The Leeds Teaching Hospitals NHS Trust - Leeds General Infirmary, Leeds
  - The Royal Wolverhampton Hospitals NHS - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rodes-Cabau J, Webb JG, Cheung A, Ye J, Dumont E, Feindel CM, Osten M, Natarajan MK, Velianou JL, Martucci G, DeVarennes B, Chisholm R, Peterson MD, Lichtenstein SV, Nietlispach F, Doyle D, DeLarochelliere R, Teoh K, Chu V, Dancea A, Lachapelle K, Cheema A, Latter D, Horlick E. Transcatheter aortic valve implantation for the treatment of severe symptomatic aortic stenosis in patients at very high or prohibitive surgical risk: acute and late outcomes of the multicenter Canadian experience. J Am Coll Cardiol. 2010 Mar 16;55(11):1080-90. doi: 10.1016/j.jacc.2009.12.014. Epub 2010 Jan 22. PMID 20096533
- [Result] Thomas M, Schymik G, Walther T, Himbert D, Lefevre T, Treede H, Eggebrecht H, Rubino P, Michev I, Lange R, Anderson WN, Wendler O. Thirty-day results of the SAPIEN aortic Bioprosthesis European Outcome (SOURCE) Registry: A European registry of transcatheter aortic valve implantation using the Edwards SAPIEN valve. Circulation. 2010 Jul 6;122(1):62-9. doi: 10.1161/CIRCULATIONAHA.109.907402. Epub 2010 Jun 21. PMID 20566953
- [Result] Lefevre T, Kappetein AP, Wolner E, Nataf P, Thomas M, Schachinger V, De Bruyne B, Eltchaninoff H, Thielmann M, Himbert D, Romano M, Serruys P, Wimmer-Greinecker G; PARTNER EU Investigator Group. One year follow-up of the multi-centre European PARTNER transcatheter heart valve study. Eur Heart J. 2011 Jan;32(2):148-57. doi: 10.1093/eurheartj/ehq427. Epub 2010 Nov 12. PMID 21075775
- [Result] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Result] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Result] Popma JJ, Adams DH, Reardon MJ, Yakubov SJ, Kleiman NS, Heimansohn D, Hermiller J Jr, Hughes GC, Harrison JK, Coselli J, Diez J, Kafi A, Schreiber T, Gleason TG, Conte J, Buchbinder M, Deeb GM, Carabello B, Serruys PW, Chenoweth S, Oh JK; CoreValve United States Clinical Investigators. Transcatheter aortic valve replacement using a self-expanding bioprosthesis in patients with severe aortic stenosis at extreme risk for surgery. J Am Coll Cardiol. 2014 May 20;63(19):1972-81. doi: 10.1016/j.jacc.2014.02.556. Epub 2014 Mar 19. PMID 24657695
- [Result] Adams DH, Popma JJ, Reardon MJ, Yakubov SJ, Coselli JS, Deeb GM, Gleason TG, Buchbinder M, Hermiller J Jr, Kleiman NS, Chetcuti S, Heiser J, Merhi W, Zorn G, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Conte J, Maini B, Mumtaz M, Chenoweth S, Oh JK; U.S. CoreValve Clinical Investigators. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 May 8;370(19):1790-8. doi: 10.1056/NEJMoa1400590. Epub 2014 Mar 29. PMID 24678937
- [Result] Webb JG, Wood DA. Current status of transcatheter aortic valve replacement. J Am Coll Cardiol. 2012 Aug 7;60(6):483-92. doi: 10.1016/j.jacc.2012.01.071. Epub 2012 Jun 27. PMID 22749306
- [Result] Genereux P, Head SJ, Wood DA, Kodali SK, Williams MR, Paradis JM, Spaziano M, Kappetein AP, Webb JG, Cribier A, Leon MB. Transcatheter aortic valve implantation 10-year anniversary: review of current evidence and clinical implications. Eur Heart J. 2012 Oct;33(19):2388-98. doi: 10.1093/eurheartj/ehs220. Epub 2012 Jul 31. PMID 22851654
- [Result] Buellesfeld L, Gerckens U, Schuler G, Bonan R, Kovac J, Serruys PW, Labinaz M, den Heijer P, Mullen M, Tymchak W, Windecker S, Mueller R, Grube E. 2-year follow-up of patients undergoing transcatheter aortic valve implantation using a self-expanding valve prosthesis. J Am Coll Cardiol. 2011 Apr 19;57(16):1650-7. doi: 10.1016/j.jacc.2010.11.044. PMID 21492762
- [Result] Ussia GP, Barbanti M, Petronio AS, Tarantini G, Ettori F, Colombo A, Violini R, Ramondo A, Santoro G, Klugmann S, Bedogni F, Maisano F, Marzocchi A, Poli A, De Carlo M, Napodano M, Fiorina C, De Marco F, Antoniucci D, de Cillis E, Capodanno D, Tamburino C; CoreValve Italian Registry Investigators. Transcatheter aortic valve implantation: 3-year outcomes of self-expanding CoreValve prosthesis. Eur Heart J. 2012 Apr;33(8):969-76. doi: 10.1093/eurheartj/ehr491. Epub 2012 Jan 12. PMID 22240494
- [Result] Walther T, Dewey T, Borger MA, Kempfert J, Linke A, Becht R, Falk V, Schuler G, Mohr FW, Mack M. Transapical aortic valve implantation: step by step. Ann Thorac Surg. 2009 Jan;87(1):276-83. doi: 10.1016/j.athoracsur.2008.08.017. PMID 19101311
- [Result] Walther T, Mollmann H, van Linden A, Kempfert J. Transcatheter aortic valve implantation transapical: step by step. Semin Thorac Cardiovasc Surg. 2011 Spring;23(1):55-61. doi: 10.1053/j.semtcvs.2011.05.006. PMID 21807300
- [Result] Lange R, Bleiziffer S, Piazza N, Mazzitelli D, Hutter A, Tassani-Prell P, Laborde JC, Bauernschmitt R. Incidence and treatment of procedural cardiovascular complications associated with trans-arterial and trans-apical interventional aortic valve implantation in 412 consecutive patients. Eur J Cardiothorac Surg. 2011 Nov;40(5):1105-13. doi: 10.1016/j.ejcts.2011.03.022. Epub 2011 Apr 22. PMID 21515069
- [Result] Miller DC, Blackstone EH, Mack MJ, Svensson LG, Kodali SK, Kapadia S, Rajeswaran J, Anderson WN, Moses JW, Tuzcu EM, Webb JG, Leon MB, Smith CR; PARTNER Trial Investigators and Patients; PARTNER Stroke Substudy Writing Group and Executive Committee. Transcatheter (TAVR) versus surgical (AVR) aortic valve replacement: occurrence, hazard, risk factors, and consequences of neurologic events in the PARTNER trial. J Thorac Cardiovasc Surg. 2012 Apr;143(4):832-843.e13. doi: 10.1016/j.jtcvs.2012.01.055. PMID 22424519
- [Result] Eggebrecht H, Schmermund A, Voigtlander T, Kahlert P, Erbel R, Mehta RH. Risk of stroke after transcatheter aortic valve implantation (TAVI): a meta-analysis of 10,037 published patients. EuroIntervention. 2012 May 15;8(1):129-38. doi: 10.4244/EIJV8I1A20. PMID 22391581
- [Result] Nuis RJ, Van Mieghem NM, Schultz CJ, Moelker A, van der Boon RM, van Geuns RJ, van der Lugt A, Serruys PW, Rodes-Cabau J, van Domburg RT, Koudstaal PJ, de Jaegere PP. Frequency and causes of stroke during or after transcatheter aortic valve implantation. Am J Cardiol. 2012 Jun 1;109(11):1637-43. doi: 10.1016/j.amjcard.2012.01.389. Epub 2012 Mar 15. PMID 22424581
- [Result] Sinning JM, Hammerstingl C, Vasa-Nicotera M, Adenauer V, Lema Cachiguango SJ, Scheer AC, Hausen S, Sedaghat A, Ghanem A, Muller C, Grube E, Nickenig G, Werner N. Aortic regurgitation index defines severity of peri-prosthetic regurgitation and predicts outcome in patients after transcatheter aortic valve implantation. J Am Coll Cardiol. 2012 Mar 27;59(13):1134-41. doi: 10.1016/j.jacc.2011.11.048. PMID 22440213
- [Result] Kodali SK, Williams MR, Smith CR, Svensson LG, Webb JG, Makkar RR, Fontana GP, Dewey TM, Thourani VH, Pichard AD, Fischbein M, Szeto WY, Lim S, Greason KL, Teirstein PS, Malaisrie SC, Douglas PS, Hahn RT, Whisenant B, Zajarias A, Wang D, Akin JJ, Anderson WN, Leon MB; PARTNER Trial Investigators. Two-year outcomes after transcatheter or surgical aortic-valve replacement. N Engl J Med. 2012 May 3;366(18):1686-95. doi: 10.1056/NEJMoa1200384. Epub 2012 Mar 26. PMID 22443479
- [Result] Tchetche D, Dumonteil N, Sauguet A, Descoutures F, Luz A, Garcia O, Soula P, Gabiache Y, Fournial G, Marcheix B, Carrie D, Fajadet J. Thirty-day outcome and vascular complications after transarterial aortic valve implantation using both Edwards Sapien and Medtronic CoreValve bioprostheses in a mixed population. EuroIntervention. 2010 Jan;5(6):659-65. doi: 10.4244/eijv5i6a109. PMID 20142215
- [Result] Van Mieghem NM, Nuis RJ, Piazza N, Apostolos T, Ligthart J, Schultz C, de Jaegere PP, Serruys PW. Vascular complications with transcatheter aortic valve implantation using the 18 Fr Medtronic CoreValve System: the Rotterdam experience. EuroIntervention. 2010 Jan;5(6):673-9. doi: 10.4244/eijv5i6a111. PMID 20142217
- [Result] Piazza N, Nuis RJ, Tzikas A, Otten A, Onuma Y, Garcia-Garcia H, Schultz C, van Domburg R, van Es GA, van Geuns R, de Jaegere P, Serruys PW. Persistent conduction abnormalities and requirements for pacemaking six months after transcatheter aortic valve implantation. EuroIntervention. 2010 Sep;6(4):475-84. doi: 10.4244/EIJ30V6I4A80. PMID 20884435
- [Result] Fraccaro C, Buja G, Tarantini G, Gasparetto V, Leoni L, Razzolini R, Corrado D, Bonato R, Basso C, Thiene G, Gerosa G, Isabella G, Iliceto S, Napodano M. Incidence, predictors, and outcome of conduction disorders after transcatheter self-expandable aortic valve implantation. Am J Cardiol. 2011 Mar 1;107(5):747-54. doi: 10.1016/j.amjcard.2010.10.054. Epub 2011 Jan 19. PMID 21247519
- [Result] van der Boon RM, Nuis RJ, Van Mieghem NM, Jordaens L, Rodes-Cabau J, van Domburg RT, Serruys PW, Anderson RH, de Jaegere PP. New conduction abnormalities after TAVI--frequency and causes. Nat Rev Cardiol. 2012 May 1;9(8):454-63. doi: 10.1038/nrcardio.2012.58. PMID 22547171
- [Result] Tzikas A, van Dalen BM, Van Mieghem NM, Gutierrez-Chico JL, Nuis RJ, Kauer F, Schultz C, Serruys PW, de Jaegere PP, Geleijnse ML. Frequency of conduction abnormalities after transcatheter aortic valve implantation with the Medtronic-CoreValve and the effect on left ventricular ejection fraction. Am J Cardiol. 2011 Jan 15;107(2):285-9. doi: 10.1016/j.amjcard.2010.09.015. Epub 2010 Dec 2. PMID 21129715
- [Result] Sherif MA, Abdel-Wahab M, Stocker B, Geist V, Richardt D, Tolg R, Richardt G. Anatomic and procedural predictors of paravalvular aortic regurgitation after implantation of the Medtronic CoreValve bioprosthesis. J Am Coll Cardiol. 2010 Nov 9;56(20):1623-9. doi: 10.1016/j.jacc.2010.06.035. PMID 21050971
- [Result] Takagi K, Latib A, Al-Lamee R, Mussardo M, Montorfano M, Maisano F, Godino C, Chieffo A, Alfieri O, Colombo A. Predictors of moderate-to-severe paravalvular aortic regurgitation immediately after CoreValve implantation and the impact of postdilatation. Catheter Cardiovasc Interv. 2011 Sep 1;78(3):432-43. doi: 10.1002/ccd.23003. Epub 2011 Jul 25. PMID 21793168
- [Derived] Manoharan G, Van Mieghem NM, Windecker S, Bosmans J, Bleiziffer S, Modine T, Linke A, Scholtz W, Chevalier B, Gooley R, Zeng C, Oh JK, Grube E. 1-Year Outcomes With the Evolut R Self-Expanding Transcatheter Aortic Valve: From the International FORWARD Study. JACC Cardiovasc Interv. 2018 Nov 26;11(22):2326-2334. doi: 10.1016/j.jcin.2018.07.032. PMID 30466832
- [Derived] Grube E, Van Mieghem NM, Bleiziffer S, Modine T, Bosmans J, Manoharan G, Linke A, Scholtz W, Tchetche D, Finkelstein A, Trillo R, Fiorina C, Walton A, Malkin CJ, Oh JK, Qiao H, Windecker S; FORWARD Study Investigators. Clinical Outcomes With a Repositionable Self-Expanding Transcatheter Aortic Valve Prosthesis: The International FORWARD Study. J Am Coll Cardiol. 2017 Aug 15;70(7):845-853. doi: 10.1016/j.jacc.2017.06.045. PMID 28797353

DOCUMENTS (4):
  • Study Protocol (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT02592369/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02592369/SAP_001.pdf
  • Informed Consent Form: Informed Consent Form (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT02592369/ICF_002.pdf
  • Informed Consent Form: Data Release Form (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT02592369/ICF_003.pdf